CLINICAL TRIAL: NCT03692208
Title: Managing Diabetes to Gain Opportunities for a More Active Life (My Diabetes GOAL)
Brief Title: Managing Diabetes to Gain Opportunities for a More Active Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB18-0425; R01DK127961-01 (NIH)
Record Dates: First submitted 2018-09-20; First posted 2018-10-02 (Actual); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Geriatrics
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients that are enrolled in the intervention arm will receive an email message via MyChart (University of Chicago patient portal) to complete an initial questionnaire. Completion of the questionnaire will be required prior to initiating risk factor tracking and opening the portal to requests for care management support. A study team member (diabetes nurse educator) will contact the patient, if requested via the survey, to initiate telephonic care management or links to additional support services. Upon completion the study, all patients will receive a post-survey via MyChart.
  Interventions: Behavioral: My Diabetes Goal Survey and Optional Care Management
- Delayed Intervention/Control (Active Comparator): Patients enrolled in the delayed intervention arm will receive usual care for the first 6 months, and then will receive the survey and intervention as stated above.
  Interventions: Behavioral: My Diabetes Goal Survey and Optional Care Management

INTERVENTIONS:
Behavioral: My Diabetes Goal Survey and Optional Care Management — The intervention is already described in the intervention arm description.

SUMMARY:
The purpose of this novel patient-facing disease management intervention is to develop and test a system embedded within the electronic medical record to engage patients in personalized goal setting and chronic disease management.

DETAILED DESCRIPTION:
The purpose of this novel patient-facing disease management intervention, My Diabetes GOAL, is to develop and test a system embedded within the electronic medical record to engage patients in personalized goal setting and chronic disease management by: 1) establishing personalized goals of care based on comorbidities and preferences, 2) tracking diabetes measures against personalized goals, and 3) selecting the route and intensity of care management to help patients achieve their goals (e.g., telephonic care management, in-person care management, and self-care resources). This application can be used to individualize care, increase engagement with patient portals, and improve patient self-efficacy, as they take a more active role in their care.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older
* Diagnosis of Type 2 Diabetes
* Enrolled in MyChart (University of Chicago Patient Portal)
* Outpatient clinic visit in the prior year

Exclusion Criteria:

* Under 64 years of age
* No type 2 diabetes
* Not enrolled in MyChart
* No outpatient clinic visit in the prior year

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elbert S Huang, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Zhu M, Cui M, Nathan AG, Press VG, Wan W, Miles C, Ali R, Pusinelli M, Huisingh-Scheetz M, Huang ES. A nurse driven care management program to engage older diabetes patients in personalized goal setting and disease management. Health Sci Rep. 2024 Jun 23;7(6):e2208. doi: 10.1002/hsr2.2208. eCollection 2024 Jun. PMID 38915356

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 110 Participants were randomized to either intervention or delayed intervention, but only 75 participants completed the initial survey immediately after randomization that was a required element to participate in the study.
Period: Overall Study
Arm/Group | Intervention | Delayed Intervention/Control
Started | 57 (randomized to arm) | 53 (randomized to arm)
Received Allocated Intervention (Received Allocated Intervention) | 42 | 33
Follow-Up Survey | 41 | 25
Completed (Excluded from final analysis: withdrawn participants) | 50 (3 participants excluded from final analysis) | 50 (7 participants excluded from final analysis)
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Population: Does not include 7 participants in the intervention arm and 3 from the delayed intervention arm who withdrew from the study prior to receiving the intervention.
Groups:
- Delayed Intervention: Patients enrolled in the delayed intervention arm will receive usual care for the first 6 months, and then will receive the survey and intervention as stated above.
- Total: Total of all reporting groups
Arm/Group | Intervention | Delayed Intervention | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.4 (5.0) | 72.7 (5.5) | 72.5 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 39 | 68
  Male | 21 | 11 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 48 | 49 | 97
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 31 | 39 | 70
  White | 17 | 8 | 25
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100
A1c [Mean (Standard Deviation); unit: % (percentage of A1c)] — Population: There are missing baseline A1C values for both study arms.
  % (percentage of A1c)
    number analyzed (Participants) | 42 | 46 | 88
    (all) | 7.1 (0.8) | 7.2 (1.3) | 7.1 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Documentation of Diabetes Goal
Description: Documentation of a personalized goal for diabetes care (e.g., A1C target) of diabetes care (yes or no).
Time Frame: Baseline, 6 months
Population: We reviewed the electronic health records to assess how many participants of the total sample of 100 participants had a documented goal in the EHR at baseline and at months.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Arm: Patients that are enrolled in the intervention arm will receive an email message via MyChart (University of Chicago patient portal) to complete an initial questionnaire. Completion of the questionnaire will be required prior to initiating risk factor tracking and opening the portal to requests for care management support. A study team member (diabetes nurse educator) will contact the patient, if requested via the survey, to initiate telephonic care management or links to additional support services. Upon completion the study, all patients will receive a post-survey via MyChart.
- Delayed Intervention Arm: Patients enrolled in the delayed intervention arm will receive usual care for the first 6 months, and then will receive the survey and intervention as stated.
Arm/Group | Intervention Arm | Delayed Intervention Arm
Number analyzed (Participants) | 50 | 50
Participants
  Baseline: Documentation of Goals | 21 | 27
  Baseline: No Documentation of Goals | 29 | 23
  6-month Trial: Documentation of Goals | 45 | 22
  6-month Trial: No Documentation of Goals | 5 | 28
Statistical Analysis 1: Comparison: Intervention Arm vs Delayed Intervention Arm; Test type: Other — Quantitative outcomes from chart and survey data were summarized by basic descriptive statistics; p < 0.01, Chi-squared — P-values were calculated. Only P values of <0.05 were considered statistically significant; Chi-squared tests, Fisher's Exact tests, two-sample t-tests, and paired two-sample t-tests were utilized to assess the outcomes between study arms

2. Secondary Outcome: Personalized A1C Goals
Description: The A1C goal outcome is based on a survey response and is distinct from the measured A1C from laboratory testing. The number of analyzed A1C goal results is therefore dependent on the number of survey respondents.
Time Frame: Baseline, 6 months
Population: The number of participants analyzed is less than 50 because of incomplete collection of personalized A1c goals at the 6 month timepoint.
Measure: Mean (Standard Deviation); unit: % (percentage A1c)
Groups:
- Delayed Intervention: Patients enrolled in the delayed intervention arm will receive usual care for the first 6 months, and then will receive the survey and intervention as stated.
Arm/Group | Intervention | Delayed Intervention
Number analyzed (Participants) | 35 | 28
% (percentage A1c)
  Baseline | 6.6 (0.7) | 6.9 (1.6)
  6 months: number analyzed (Participants) | 34 | 24
  6 months | 7.0 (0.9) | 6.7 (0.6)

3. Secondary Outcome: Patient Ability to Reach Personalized Goals
Description: Using EHR data, we will measure whether or not patients are reaching the goals they have documented in the survey.
Time Frame: Baseline, 6 month
Population: We reviewed the electronic health records to assess how many participants of the Intervention Arm reached their documented goals at baseline and at 6 months. The denominator is limited to participants with survey responses and lab values.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Delayed Intervention/Control
Number analyzed (Participants) | 32 | 25
Participants
  Baseline: Achieved Goal | 10 | 10
  Baseline: Goal not achieved | 22 | 15
  6 month trial: number analyzed (Participants) | 30 | 17
  6 month trial: Achieved Goal | 13 | 5
  6 month trial: Goal not achieved | 17 | 12

4. Other Pre Specified Outcome: Health Care Utilization
Description: We will utilize the EHR to determine the frequency of referrals to telephone care management, the source of referrals (population management, physician), the patient predictors of referrals, and to characterize frequency and content of telephonic management.
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed. The data collection period was 23 months.
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Groups:
- Intervention Arm: Experimental: Intervention Patients that are enrolled in the intervention arm will receive an email message via MyChart (University of Chicago patient portal) to complete an initial questionnaire. Completion of the questionnaire will be required prior to initiating risk factor tracking and opening the portal to requests for care management support. A study team member (diabetes nurse educator) will contact the patient, if requested via the survey, to initiate telephonic care management or links to additional support services. Upon completion the study, all patients will receive a post-survey via MyChart.
Arm/Group | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/08/NCT03692208/Prot_SAP_000.pdf